CLINICAL TRIAL: NCT02304458
Title: A Phase 1/2 Study of Nivolumab in Children, Adolescents, and Young Adults With Recurrent or Refractory Solid Tumors as a Single Agent and in Combination With Ipilimumab
Brief Title: Nivolumab With or Without Ipilimumab in Treating Younger Patients With Recurrent or Refractory Solid Tumors or Sarcomas
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-01222; NCI-2014-01222 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ADVL1412 (Other: Pediatric Early Phase Clinical Trial Network); ADVL1412 (Other: CTEP); UM1CA097452 (NIH)
Record Dates: First submitted 2014-11-26; First posted 2014-12-02 (Estimated); Results first posted 2023-01-10 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-09

CONDITIONS: Metastatic Melanoma; Recurrent Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor; Recurrent Hodgkin Lymphoma; Recurrent Malignant Solid Neoplasm; Recurrent Melanoma; Recurrent Neuroblastoma; Recurrent Non-Hodgkin Lymphoma; Recurrent Osteosarcoma; Recurrent Rhabdomyosarcoma; Refractory Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor; Refractory Hodgkin Lymphoma; Refractory Malignant Solid Neoplasm; Refractory Melanoma; Refractory Neuroblastoma; Refractory Non-Hodgkin Lymphoma; Refractory Osteosarcoma; Refractory Rhabdomyosarcoma; Stage III Cutaneous Melanoma AJCC v7; Stage IIIA Cutaneous Melanoma AJCC v7; Stage IIIB Cutaneous Melanoma AJCC v7; Stage IIIC Cutaneous Melanoma AJCC v7; Stage IV Cutaneous Melanoma AJCC v6 and v7; Unresectable Melanoma
MeSH Terms: conditions — Melanoma; Neuroectodermal Tumors, Primitive, Peripheral; Hodgkin Disease; Neuroblastoma; Lymphoma, Non-Hodgkin; Osteosarcoma; Rhabdomyosarcoma | interventions — Ipilimumab; CTLA-4 Antigen; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (nivolumab, ipilimumab) (Experimental): See Detailed Description
  Interventions: Biological: Ipilimumab; Other: Laboratory Biomarker Analysis; Biological: Nivolumab; Other: Pharmacological Study

INTERVENTIONS:
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; Ipilimumab Biosimilar CS1002; MDX-010; MDX-CTLA4; Yervoy
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; CMAB819; MDX-1106; NIVO; Nivolumab Biosimilar CMAB819; ONO-4538; Opdivo
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I/II trial studies the side effects and best dose of nivolumab when given with or without ipilimumab to see how well they work in treating younger patients with solid tumors or sarcomas that have come back (recurrent) or do not respond to treatment (refractory). Immunotherapy with monoclonal antibodies, such as nivolumab and ipilimumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. It is not yet known whether nivolumab works better alone or with ipilimumab in treating patients with recurrent or refractory solid tumors or sarcomas.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the tolerability, and define and describe the toxicities of nivolumab administered as a single agent in children with relapsed or refractory solid tumors at the adult recommended dose of 3 mg/kg.

II. Determine if systemic nivolumab exposure in children is similar to the systemic exposure in adults following a 3 mg/kg dose.

III. Determine the maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D) and define and describe the toxicities of nivolumab plus ipilimumab administered to children with relapsed or refractory solid tumors.

IV. Assess antitumor effects of nivolumab across selected childhood solid tumors in seven expansion cohorts (Parts B1-B6, B8); neuroblastoma (2 cohorts: measurable disease, metaiodobenzylguanidine [MIBG] positive only non-measurable disease), osteosarcoma, rhabdomyosarcoma, Ewing sarcoma, Hodgkin lymphoma, and non-Hodgkin lymphoma.

V. Assess antitumor effects of nivolumab in combination with ipilimumab across selected childhood solid tumors in two dose combinations (Part D and Part E).

VI. Characterize the pharmacokinetics of nivolumab alone and in combination with ipilimumab, including area under the curve (AUC), concentration maximum (Cmax), concentration minimum (Cmin), using intensive sampling.

VII. Assess immunogenicity of nivolumab alone and in combination with ipilimumab by measuring anti-drug antibody (ADA) levels.

SECONDARY OBJECTIVES:

I. Conduct exploratory studies of the phenotypic and functional effects of nivolumab (alone and in combination with ipilimumab), as well as changes in antibodies to previously vaccinated viruses, in serum samples.

II. Explore whether correlations exist between PD-L1 expression on tumor and antitumor effects of nivolumab (alone and in combination with ipilimumab) in pediatric solid tumors and to conduct exploratory studies of potential tumor associated biomarkers of response in tumor tissue (at least five out of the following markers: NRAS, BRAF, MEK, KIT, PDGF, TP53, RB1 and BRCA1, Akt phosphorylation, IL-17 or PD-L1).

III. Explore presence of tumor infiltrating lymphocytes and their association with antitumor effects of nivolumab (alone and in combination with ipilimumab).

IV. Conduct exploratory studies of the effect of nivolumab (alone or in combination with ipilimumab) on cytokine levels in serum samples.

V. For Part E, determine tumor mutational burden of diagnostic specimens using FoundationOneCDx testing to explore immune- related gene expression or mutation and its association with antitumor response to nivolumab in combination with ipilimumab.

OUTLINE: This is a phase I, dose-escalation study of nivolumab followed by a phase II study.

PART A (COMPLETED): Patients with recurrent or refractory solid tumors receive nivolumab intravenously (IV) over 30 minutes on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

PART B (COMPLETED): Patients with neuroblastoma, osteosarcoma, rhabdomyosarcoma, Ewing sarcoma, Hodgkin lymphoma, non-Hodgkin lymphoma, or melanoma receive nivolumab as in Part A.

PART C (COMPLETED):

INDUCTION: Patients receive nivolumab IV over 60 minutes and ipilimumab IV over 90 minutes on day 1. Treatment repeats every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Patients receive nivolumab IV as in Part A. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

PART D (COMPLETED):

INDUCTION: Patients with neuroblastoma, osteosarcoma, rhabdomyosarcoma, Ewing sarcoma, Hodgkin lymphoma, non-Hodgkin lymphoma, or melanoma receive nivolumab IV and ipilimumab IV as in Part C. Treatment repeats every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity.

MAINTENANCE: Patients receive nivolumab IV over 30 minutes on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

PART E: Patients receive nivolumab IV over 30 minutes on day 1 and ipilimumab IV over 90 minutes on day 1. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive nivolumab IV over 30 minutes on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at approximately 100 days, every 6 months for up to 24 months, and then annually for up to 60 months.

ELIGIBILITY:
Inclusion Criteria:

* Parts A & C: patients must be >= 12 months and < 18 years of age at the time of study enrollment
* Parts B1-B6, B8, D1-D6, E3, E4: patients must be >= 12 months and =< 30 years of age at the time of study enrollment
* Part B7: patients must be >= 12 months and < 18 years of age at the time of study enrollment
* Patients must have had histologic verification of malignancy at original diagnosis or relapse

  * Parts A & C: patients with recurrent or refractory solid tumors, without central nervous system (CNS) tumors or known CNS metastases, are eligible; note: CNS imaging for patients without a known history of CNS disease is only required if clinically indicated
  * Part B1: patients with relapsed or refractory neuroblastoma
  * Part B2: patients with relapsed or refractory osteosarcoma
  * Part B3: patients with relapsed or refractory rhabdomyosarcoma
  * Part B4: patients with relapsed or refractory Ewing sarcoma or peripheral primitive neuroectodermal tumor (PNET)
  * Part B5: patients with relapsed or refractory Hodgkin lymphoma
  * Part B6: patients with relapsed or refractory non-Hodgkin lymphoma
  * Part B7: patients with unresectable melanoma or metastatic melanoma or relapsed melanoma or refractory melanoma
  * Part B8: Patients with relapsed or refractory neuroblastoma (MIBG evaluable disease without Response Evaluation Criteria in Solid Tumors [RECIST] measurable lesion)
  * Once the dose-escalation portion of Part A is completed, cohorts that are open concurrently for eligible patients (including Parts B and C and potential pharmacokinetic [PK] expansion cohorts) may be selected at the treating physician's discretion pending slot availability; in the event a disease group cohort in Part B is completed after the initial stage of Simon's optimal two-stage design, for selected disease cohorts, a corresponding cohort in the same disease group for select disease types will be open in Part D:
  * Part D1: Patients with relapsed or refractory neuroblastoma
  * Part D2: Patients with relapsed or refractory osteosarcoma
  * Part D3: Patients with relapsed or refractory rhabdomyosarcoma
  * Part D4: Patients with relapsed or refractory Ewing sarcoma or peripheral PNET
  * Part D5: Patients with relapsed or refractory non-Hodgkin lymphoma
  * Part D6: Patients with relapsed or refractory neuroblastoma (MIBG evaluable disease without RECIST measurable lesion)
  * Part E3: Patients with relapsed or refractory rhabdomyosarcoma
  * Part E4: Patients with relapsed or refractory Ewing sarcoma or peripheral PNET
* Parts A & C: patients must have either measurable or evaluable disease
* Parts B, D & E: patients must have measurable disease for Parts B1-B6, D1-D5, E3 and E4; melanoma patients in Part B7 must have either measurable or evaluable disease; neuroblastoma patients in Parts B8 and D6 must be evaluable for MIBG response without evidence of RECIST measurable lesions
* Patient's current disease state must be one for which there is no known curative therapy or therapy proven to prolong survival with an acceptable quality of life
* Karnofsky >= 50% for patients > 16 years of age and Lansky >= 60 for patients =< 16 years of age; patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Patients must have fully recovered from the acute toxic effects of all prior anti-cancer therapy and must meet the following minimum duration from prior anti-cancer directed therapy prior to enrollment; if after the required timeframe, the defined eligibility criteria are met, e.g. blood count criteria, the patient is considered to have recovered adequately

  * Cytotoxic chemotherapy or other anti-cancer agents known to be myelosuppressive

    * At least 21 days after the last dose of cytotoxic or myelosuppressive chemotherapy (42 days if prior nitrosourea)
  * Hematopoietic growth factors: At least 14 days after the last dose of a long-acting growth factor (e.g. pegfilgrastim) or 7 days for short-acting growth factor; for agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur; the duration of this interval must be discussed with the study chair
  * Anti-cancer agents not known to be myelosuppressive (e.g. not associated with reduced platelet or absolute neutrophil count [ANC] counts): At least 7 days after the last dose of agent
  * Interleukins, interferons and cytokines (other than hematopoietic growth factors): >= 21 days after the completion of interleukins, interferon or cytokines (other than hematopoietic growth factors)
  * Antibodies: >= 21 days must have elapsed from infusion of last dose of antibody, and toxicity related to prior antibody therapy must be recovered to grade =< 1
  * External beam radiation therapy (XRT)/external beam irradiation including protons: >= 14 days after local XRT; >= 150 days after total body irradiation (TBI), craniospinal XRT or if radiation to >= 50% of the pelvis; >= 42 days if other substantial bone marrow (BM) radiation.
  * Radiopharmaceutical therapy (e.g., radiolabeled antibody, 131I-MIBG): >= 42 days must have elapsed since systemically administered radiopharmaceutical therapy
  * Cellular therapy: >= 42 days must have elapsed since the completion of any type of cellular therapy (e.g. modified T cells, natural killer [NK] cells, dendritic cells, etc.)
  * Patients must not have received prior exposure to nivolumab; for patients enrolled in Parts C, D, and E patients must not have received prior nivolumab or ipilimumab
* For patients with solid tumors without known bone marrow involvement:
* Peripheral absolute neutrophil count (ANC) >= 750/mm^3
* Platelet count >= 75,000/mm^3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment)
* Patients with known bone marrow metastatic disease will be eligible for study provided they meet the blood counts above (may receive transfusions provided they are not known to be refractory to red cell or platelet transfusions); these patients will not be evaluable for hematologic toxicity; at least 5 of every cohort of 6 patients with a solid tumor must be evaluable for hematologic toxicity, for Parts A and C; if dose-limiting hematologic toxicity is observed on either Part A or C, all subsequent patients enrolled must be evaluable for hematologic toxicity on that Part
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 ml/min/1.73 m^2 or a serum creatinine based on age/gender as follows:

  * Age 1 to < 2 years: maximum serum creatinine (mg/dL) 0.6 for males and females
  * Age 2 to < 6 years: 0.8 for males and females
  * Age 6 to < 10 years: 1 for males and females
  * Age 10 to < 13 years: 1.2 for males and females
  * Age 13 to < 16 years: 1.5 for males and 1.4 for females
  * Age >= 16 years: 1.7 for males and 1.4 for females
* Bilirubin (sum of conjugated + unconjugated) =< 1.5 x upper limit of normal (ULN) for age
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 135 U/L; for the purpose of this study, the ULN for SGPT is 45 U/L
* No evidence of dyspnea at rest, no exercise intolerance due to pulmonary insufficiency, and a pulse oximetry > 92% while breathing room air
* Serum lipase =< ULN at baseline; patients with glucose intolerance should be on a stable regimen and be monitored
* All patients and/or their parents or legally authorized representatives must sign a written informed consent; assent, when appropriate, will be obtained according to institutional guidelines
* Tissue blocks or slides must be sent for all patients; if tissue blocks or slides are unavailable, the study chair must be notified prior to enrollment

Exclusion Criteria:

* Pregnant or breast-feeding women will not be entered on this study due to risks of fetal and teratogenic adverse events as there is yet no available information regarding human fetal or teratogenic toxicities; pregnancy tests must be obtained in girls who are post-menarchal; women of childbearing potential (WOCBP) receiving nivolumab will be instructed to adhere to contraception for a period of 5 months after the last dose of nivolumab; men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 7 months after the last dose of nivolumab
* Patients requiring daily systemic corticosteroids are not eligible; patients must not have received systemic corticosteroids within 7 days prior to enrollment; if used to modify immune adverse events related to prior therapy, >= 14 days must have elapsed since last dose of corticosteroid; Note: use of topical or inhaled corticosteroids will not render a patient ineligible
* Patients who are currently receiving another investigational drug are not eligible
* Patients who are currently receiving other anti-cancer agents are not eligible
* Patients with CNS tumors or known CNS metastases will be excluded from this trial; patients with a history of CNS metastases that have been previously treated may enroll if sequential imaging shows not evidence for active disease; patients with extra axial disease (e.g. skull [bone] metastasis that do not invade the dura) may enroll if there is no evidence for CNS edema associated with the lesion
* Patients with a history of any grade autoimmune disorder are not eligible; asymptomatic laboratory abnormalities (e.g. antinuclear antibody [ANA], rheumatoid factor, altered thyroid function studies) will not render a patient ineligible in the absence of a diagnosis of an autoimmune disorder
* Patients with >= grade 2 hypothyroidism due to history of autoimmunity are not eligible; note: hypothyroidism due to previous irradiation on thyroidectomy will not impact eligibility
* Patients who have an uncontrolled infection are not eligible
* Patients with a history of congestive heart failure (CHF) or are at risk because of underlying cardiovascular disease or exposure to cardiotoxic drugs must have adequate cardiac function as clinically indicated:

  * Corrected QT interval (QTC) =< 480 msec
  * Shortening fraction of >= 27% by echocardiogram or ejection fraction of >= 50% by gated radionuclide study
* Patients with known human immunodeficiency virus (HIV) or hepatitis B or C are excluded
* Patients who have received prior solid organ transplantation are not eligible
* Patient who have received allotransplantation are not eligible
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible
* Patients who have received prior anti-PD1 directed therapy (monoclonal antibody [mAb] or small molecule) are not eligible
* Parts C, D, and E: patients who have received prior ipilimumab are not eligible

Ages: 12 Months to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 140 (Actual)
Dates: Start 2015-03-30 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2023-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Crystal L Mackall, Principal Investigator — COG Phase I Consortium
Locations (25):
- United States (24):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Davis KL, Fox E, Merchant MS, Reid JM, Kudgus RA, Liu X, Minard CG, Voss S, Berg SL, Weigel BJ, Mackall CL. Nivolumab in children and young adults with relapsed or refractory solid tumours or lymphoma (ADVL1412): a multicentre, open-label, single-arm, phase 1-2 trial. Lancet Oncol. 2020 Apr;21(4):541-550. doi: 10.1016/S1470-2045(20)30023-1. Epub 2020 Mar 17. PMID 32192573
- [Derived] Hattinger CM, Patrizio MP, Magagnoli F, Luppi S, Serra M. An update on emerging drugs in osteosarcoma: towards tailored therapies? Expert Opin Emerg Drugs. 2019 Sep;24(3):153-171. doi: 10.1080/14728214.2019.1654455. Epub 2019 Aug 14. PMID 31401903

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A: 3 mg/kg Nivolumab; Part C: 1mg/kg Nivolumab and 1mg/kg Ipilimumab; Part C: 3mg/kg Nivolumab and 1mg/kg Ipilimumab; Part C PK: 3mg/kg Nivolumab and 1mg/kg Ipilimumab: Phase 1: Patients with solid tumors, excluding brain and CNS tumors
- Part A PK: 3 mg/kg Nivolumab: Phase 1: Patients with solid tumors, excluding brain and CNS tumors receive
- Part B: 3 mg/kg Nivolumab: Patients with relapsed or refractory neuroblastoma, osteosarcoma, rhabdomyosarcoma, Ewing Sarcoma or Peripheral PNET, Hodgkin Lymphoma, Non-Hodgkin Lymphoma, unresectable melanoma or metastatic melanoma or relapsed melanoma or refractory melanoma, neuroblastoma (MIBG evaluable without RECIST evaluable disease)
- Part D: 3mg/kg Nivolumab and 1mg/kg Ipilimumab: Patients with relapsed or refractory osteosarcoma, rhabdomyosarcoma, Ewing Sarcoma or Peripheral PNET
- Part E: 1mg/kg Nivolumab and 3mg/kg Ipilimumab: Patients with relapsed or refractory rhabdomyosarcoma, Ewing Sarcoma, or Peripheral PNET
Period: Overall Study
Arm/Group | Part A: 3 mg/kg Nivolumab | Part A PK: 3 mg/kg Nivolumab | Part B: 3 mg/kg Nivolumab | Part C: 1mg/kg Nivolumab and 1mg/kg Ipilimumab | Part C: 3mg/kg Nivolumab and 1mg/kg Ipilimumab | Part C PK: 3mg/kg Nivolumab and 1mg/kg Ipilimumab | Part D: 3mg/kg Nivolumab and 1mg/kg Ipilimumab | Part E: 1mg/kg Nivolumab and 3mg/kg Ipilimumab
Started | 7 | 6 | 72 | 6 | 6 | 6 | 29 | 8
Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not Completed | 7 | 6 | 71 | 6 | 6 | 6 | 29 | 8
Not completed — Adverse Event | 0 | 0 | 7 | 0 | 0 | 0 | 3 | 4
Not completed — Death | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 4 | 6 | 38 | 5 | 6 | 6 | 21 | 4
Not completed — Physician Decision | 2 | 0 | 16 | 1 | 0 | 0 | 3 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 7 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: 3 mg/kg Nivolumab | Part A PK: 3 mg/kg Nivolumab | Part B: 3 mg/kg Nivolumab | Part C: 1mg/kg Nivolumab and 1mg/kg Ipilimumab | Part C: 3mg/kg Nivolumab and 1mg/kg Ipilimumab | Part C PK: 3mg/kg Nivolumab and 1mg/kg Ipilimumab | Part D: 3mg/kg Nivolumab and 1mg/kg Ipilimumab | Part E: 1mg/kg Nivolumab and 3mg/kg Ipilimumab | Total
Number analyzed (Participants) | 7 | 6 | 72 | 6 | 6 | 6 | 29 | 8 | 140
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 6 | 59 | 6 | 6 | 6 | 18 | 4 | 112
  Between 18 and 65 years | 0 | 0 | 13 | 0 | 0 | 0 | 11 | 4 | 28
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 12 [5 to 13] | 9.5 [7 to 15] | 15 [1 to 27] | 15 [12 to 15] | 14.5 [11 to 17] | 8.5 [4 to 27] | 17 [5 to 27] | 19 [11 to 28] | 15 [1 to 28]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 28 | 1 | 3 | 4 | 8 | 5 | 55
  Male | 2 | 5 | 44 | 5 | 3 | 2 | 21 | 3 | 85
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 9 | 1 | 1 | 1 | 5 | 1 | 21
  Not Hispanic or Latino | 5 | 5 | 62 | 5 | 5 | 5 | 23 | 7 | 117
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 5 | 1 | 1 | 0 | 0 | 0 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 8 | 1 | 1 | 0 | 2 | 0 | 12
  White | 7 | 6 | 51 | 3 | 4 | 4 | 23 | 8 | 106
  More than one race | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 6 | 1 | 0 | 1 | 4 | 0 | 12

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Dose Limiting Toxicities of Nivolumab as a Single Agent or in Combination With Ipilimumab
Description: The frequency (%) of patients experiencing a dose limiting toxicity at least possibly attributable to nivolumab as a single agent or in combination with ipilimumab by study part and dose level.
Time Frame: 28 days
Population: All Eligible patients
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: 3 mg/kg Nivolumab | Part A PK: 3 mg/kg Nivolumab | Part B: 3 mg/kg Nivolumab | Part C: 1mg/kg Nivolumab and 1mg/kg Ipilimumab | Part C: 3mg/kg Nivolumab and 1mg/kg Ipilimumab | Part C PK: 3mg/kg Nivolumab and 1mg/kg Ipilimumab | Part D: 3mg/kg Nivolumab and 1mg/kg Ipilimumab | Part E: 1mg/kg Nivolumab and 3mg/kg Ipilimumab
Number analyzed (Participants) | 7 | 6 | 72 | 6 | 6 | 6 | 29 | 8
Participants | 0 | 0 | 5 | 0 | 0 | 1 | 1 | 1
Statistical Analysis 1: Comparison: Part A: 3 mg/kg Nivolumab vs Part A PK: 3 mg/kg Nivolumab vs Part B: 3 mg/kg Nivolumab vs Part C: 1mg/kg Nivolumab and 1mg/kg Ipilimumab vs Part C: 3mg/kg Nivolumab and 1mg/kg Ipilimumab vs Part C PK: 3mg/kg Nivolumab and 1mg/kg Ipilimumab vs Part D: 3mg/kg Nivolumab and 1mg/kg Ipilimumab vs Part E: 1mg/kg Nivolumab and 3mg/kg Ipilimumab; Test type: Other — Maximum Tolerate Dose Level was determined by the rolling-6 design; Maximum Tolerate Dose Level = 3 — Maximum Tolerate Dose Level is 3 mg/kg Nivolumab

2. Primary Outcome: Antitumor Effect of Nivolumab as a Single Agent or in Combination With Ipilimumab
Description: Frequency of disease response (best overall response of partial or complete response) assessed per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR by study part and dose level.
Time Frame: Up to 5 years
Population: All Eligible patients
Measure: Count of Participants; unit: Participants
Groups:
- Part B1: 3 mg/kg Nivolumab: Patients with relapsed or refractory neuroblastoma
- Part B2: 3 mg/kg Nivolumab; Part D2: 3mg/kg Nivolumab and 1mg/kg Ipilimumab: Patients with relapsed or refractory osteosarcoma
- Part B3: 3 mg/kg Nivolumab; Part D3: 3mg/kg Nivolumab and 1mg/kg Ipilimumab; Part E3: 1mg/kg Nivolumab and 3mg/kg Ipilimumab: Patients with relapsed or refractory rhabdomyosarcoma
- Part B4: 3 mg/kg Nivolumab; Part D4: 3mg/kg Nivolumab and 1mg/kg Ipilimumab: Patients with relapsed or refractory Ewing Sarcoma or Peripheral PNET
- Part B5: 3 mg/kg Nivolumab: Patients with relapsed or refractory Hodgkin Lymphoma
- Part B6: 3 mg/kg Nivolumab: Patients with relapsed or refractory Non-Hodgkin Lymphoma
- Part B7: 3 mg/kg Nivolumab: Patients with unresectable melanoma or metastatic melanoma or relapsed melanoma or refractory melanoma
- Part B8: 3 mg/kg Nivolumab: Patients with relapsed or refractory neuroblastoma (MIBG evaluable without RECIST evaluable disease)
- Part E4: 1mg/kg Nivolumab and 3mg/kg Ipilimumab: Patients with relapsed or refractory Ewing Sarcoma, or Peripheral PNET
Arm/Group | Part A: 3 mg/kg Nivolumab | Part A PK: 3 mg/kg Nivolumab | Part B1: 3 mg/kg Nivolumab | Part B2: 3 mg/kg Nivolumab | Part B3: 3 mg/kg Nivolumab | Part B4: 3 mg/kg Nivolumab | Part B5: 3 mg/kg Nivolumab | Part B6: 3 mg/kg Nivolumab | Part B7: 3 mg/kg Nivolumab | Part B8: 3 mg/kg Nivolumab | Part C: 1mg/kg Nivolumab and 1mg/kg Ipilimumab | Part C: 3mg/kg Nivolumab and 1mg/kg Ipilimumab | Part C PK: 3mg/kg Nivolumab and 1mg/kg Ipilimumab | Part D2: 3mg/kg Nivolumab and 1mg/kg Ipilimumab | Part D3: 3mg/kg Nivolumab and 1mg/kg Ipilimumab | Part D4: 3mg/kg Nivolumab and 1mg/kg Ipilimumab | Part E3: 1mg/kg Nivolumab and 3mg/kg Ipilimumab | Part E4: 1mg/kg Nivolumab and 3mg/kg Ipilimumab
Number analyzed (Participants) | 7 | 6 | 10 | 10 | 11 | 10 | 12 | 10 | 1 | 8 | 6 | 6 | 6 | 10 | 10 | 9 | 5 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0

3. Secondary Outcome: Pharmacodynamics of Nivolumab as a Single Agent or in Combination With Ipilimumab
Description: Median (min,max) concentration by protein, study part, and dose level.
Time Frame: Up to 28 days
Population: Data were not and will never be collected
Arm/Group | Part A: 3 mg/kg Nivolumab | Part A PK: 3 mg/kg Nivolumab | Part B: 3 mg/kg Nivolumab | Part C: 1mg/kg Nivolumab and 1mg/kg Ipilimumab | Part C: 3mg/kg Nivolumab and 1mg/kg Ipilimumab | Part C PK: 3mg/kg Nivolumab and 1mg/kg Ipilimumab | Part D: 3mg/kg Nivolumab and 1mg/kg Ipilimumab | Part E: 1mg/kg Nivolumab and 3mg/kg Ipilimumab
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Area Under the Drug Concentration Curve of Nivolumab as a Single Agent or in Combination With Ipilimumab
Description: The median (min,max) of the area under the drug concentration curve for nivolumab as a single agent or in combination with ipilimumab by study part and dose level. Measured during cycle 1 at 0, 24,72,192, and 360 hours post-dose.
Time Frame: Up to 15 days
Population: All eligible patients with data collected. Data not collected for Parts C, D, and E
Measure: Median (Full Range); unit: hr*ug/mL
Arm/Group | Part A: 3 mg/kg Nivolumab | Part A PK: 3 mg/kg Nivolumab | Part B: 3 mg/kg Nivolumab
Number analyzed (Participants) | 6 | 6 | 63
hr*ug/mL | 20744.5 [11840.0 to 31067.0] | 18338 [9383.0 to 31188.0] | 20816 [6442.0 to 133556.0]

5. Secondary Outcome: Half-life of Nivolumab as a Single Agent or in Combination With Ipilimumab
Description: The median (min,max) of the half-life of nivolumab as a single agent or in combination with ipilimumab by study part and dose level. Measured during cycle 1 at 0, 24, 72, 192, and 360 hours post-dose. The reported half-life was calculated using a linear regression of the log (concentration) versus time data for days 4, 8 and 15.
Time Frame: Up to 15 days
Population: All eligible patients with data collected. Data not collected for Parts C, D, and E
Measure: Median (Full Range); unit: hours
Arm/Group | Part A: 3 mg/kg Nivolumab | Part A PK: 3 mg/kg Nivolumab | Part B: 3 mg/kg Nivolumab
Number analyzed (Participants) | 6 | 6 | 63
hours | 312.5 [154.0 to 444.0] | 281.5 [263.0 to 426.0] | 379 [92.0 to 2772.0]

6. Secondary Outcome: Maximum Serum Concentration of Nivolumab as a Single Agent or in Combination With Ipilimumab
Description: Median (min,max) of the maximum serum concentration of nivolumab as a single agent or in combination with ipilimumab by study part and dose level. Measured during cycle 1 at 0, 24, 72, 192, and 360 hours post-dose.
Time Frame: Up to 15 days
Population: All eligible patients with data collected
Measure: Median (Full Range); unit: ug/mL
Arm/Group | Part A: 3 mg/kg Nivolumab | Part A PK: 3 mg/kg Nivolumab | Part B: 3 mg/kg Nivolumab | Part C: 1mg/kg Nivolumab and 1mg/kg Ipilimumab | Part C: 3mg/kg Nivolumab and 1mg/kg Ipilimumab | Part C PK: 3mg/kg Nivolumab and 1mg/kg Ipilimumab | Part D: 3mg/kg Nivolumab and 1mg/kg Ipilimumab | Part E: 1mg/kg Nivolumab and 3mg/kg Ipilimumab
Number analyzed (Participants) | 6 | 6 | 65 | 6 | 5 | 6 | 28 | 4
ug/mL | 80.9 [56.9 to 119.4] | 72 [39.0 to 93.7] | 68.1 [37.6 to 224.9] | 17.3 [14.4 to 23.1] | 43.3 [35.4 to 48.6] | 41.7 [23.2 to 74.4] | 34.6 [15.9 to 61.7] | 49.1 [10.0 to 62.5]

7. Secondary Outcome: Minimum Serum Concentration of Nivolumab as a Single Agent or in Combination With Ipilimumab
Description: Median (min,max) of the minimum serum concentration of nivolumab as a single agent or in combination with ipilimumab by study part and dose level. Measured during cycle 1 at 0, 24, 72, 192, and 360 hours post-dose.
Time Frame: Up to 15 days
Population: All eligible patients with data collected
Measure: Median (Full Range); unit: ug/mL
Arm/Group | Part A: 3 mg/kg Nivolumab | Part A PK: 3 mg/kg Nivolumab | Part B: 3 mg/kg Nivolumab | Part C: 1mg/kg Nivolumab and 1mg/kg Ipilimumab | Part C: 3mg/kg Nivolumab and 1mg/kg Ipilimumab | Part C PK: 3mg/kg Nivolumab and 1mg/kg Ipilimumab | Part D: 3mg/kg Nivolumab and 1mg/kg Ipilimumab | Part E: 1mg/kg Nivolumab and 3mg/kg Ipilimumab
Number analyzed (Participants) | 6 | 6 | 65 | 2 | 5 | 4 | 23 | 3
ug/mL | 29.6 [13.7 to 60.9] | 30.4 [9.7 to 46.7] | 26.4 [8.9 to 85.3] | 3.8 [2.0 to 5.6] | 10.5 [7.4 to 14.0] | 9.2 [7.9 to 12.9] | 10.8 [2.9 to 30.0] | 8 [7.7 to 12.8]

8. Secondary Outcome: Clearance of Nivolumab as a Single Agent or in Combination With Ipilimumab
Description: Median (min,max) of the clearance of nivolumab as a single agent or in combination with ipilimumab by study part and dose level. Measured during cycle 1 at 0, 24, 72, 192, and 360 hours post-dose.
Time Frame: Up to 15 days
Population: All eligible patients with data collected. Data not collected for Parts C, D, and E
Measure: Median (Full Range); unit: mL/hr/kg
Arm/Group | Part A: 3 mg/kg Nivolumab | Part A PK: 3 mg/kg Nivolumab | Part B: 3 mg/kg Nivolumab
Number analyzed (Participants) | 6 | 6 | 63
mL/hr/kg | 0.1 [0.1 to 0.3] | 0.2 [0.1 to 0.3] | 0.1 [0.0 to 0.5]

9. Secondary Outcome: PD-L1 Expression of Nivolumab as a Single Agent or in Combination With Ipilimumab
Description: Median (min, max) of PD-L1 expression levels by study part, dose level, and disease cohort.
Time Frame: Cycle 1 (21 days)
Population: All Eligible patients
Measure: Median (Full Range); unit: percent
Arm/Group | Part A: 3 mg/kg Nivolumab | Part A PK: 3 mg/kg Nivolumab | Part B1: 3 mg/kg Nivolumab | Part B2: 3 mg/kg Nivolumab | Part B3: 3 mg/kg Nivolumab | Part B4: 3 mg/kg Nivolumab | Part B5: 3 mg/kg Nivolumab | Part B6: 3 mg/kg Nivolumab | Part B7: 3 mg/kg Nivolumab | Part B8: 3 mg/kg Nivolumab | Part C: 1mg/kg Nivolumab and 1mg/kg Ipilimumab | Part C: 3mg/kg Nivolumab and 1mg/kg Ipilimumab | Part C PK: 3mg/kg Nivolumab and 1mg/kg Ipilimumab | Part D2: 3mg/kg Nivolumab and 1mg/kg Ipilimumab | Part D3: 3mg/kg Nivolumab and 1mg/kg Ipilimumab | Part D4: 3mg/kg Nivolumab and 1mg/kg Ipilimumab | Part E3: 1mg/kg Nivolumab and 3mg/kg Ipilimumab | Part E4: 1mg/kg Nivolumab and 3mg/kg Ipilimumab
Number analyzed (Participants) | 7 | 6 | 10 | 10 | 11 | 10 | 12 | 10 | 1 | 8 | 6 | 6 | 6 | 10 | 10 | 9 | 5 | 3
percent | 0 [0.0 to 0.0] | 0 [0.0 to 0.0] | 2.5 [0.0 to 70.0] | 0 [0.0 to 1.0] | 0 [0.0 to 3.0] | 0 [0.0 to 1.0] | 100 [30.0 to 100.0] | 7.5 [0.0 to 100.0] | 0 [0.0 to 0.0] | 0 [0.0 to 0.0] | 0 [0.0 to 97.0] | 3 [0.0 to 100.0] | 0 [0.0 to 0.0] | 0 [0.0 to 0.0] | 0 [0.0 to 3.0] | 0 [0.0 to 25.0] | 0 [0.0 to 0.0] | 0 [0.0 to 0.0]

10. Secondary Outcome: Biomarker Expression Analysis of Nivolumab as a Single Agent or in Combination With Ipilimumab
Description: Median (min, max) expression levels by biomarker, dose level, study part, and disease cohort.
Time Frame: Cycle 1 (21 days)
Population: Data were not and will never be collected
Arm/Group | Part A: 3 mg/kg Nivolumab | Part A PK: 3 mg/kg Nivolumab | Part B1: 3 mg/kg Nivolumab | Part B2: 3 mg/kg Nivolumab | Part B3: 3 mg/kg Nivolumab | Part B4: 3 mg/kg Nivolumab | Part B5: 3 mg/kg Nivolumab | Part B6: 3 mg/kg Nivolumab | Part B7: 3 mg/kg Nivolumab | Part B8: 3 mg/kg Nivolumab | Part C: 1mg/kg Nivolumab and 1mg/kg Ipilimumab | Part C: 3mg/kg Nivolumab and 1mg/kg Ipilimumab | Part C PK: 3mg/kg Nivolumab and 1mg/kg Ipilimumab | Part D2: 3mg/kg Nivolumab and 1mg/kg Ipilimumab | Part D3: 3mg/kg Nivolumab and 1mg/kg Ipilimumab | Part D4: 3mg/kg Nivolumab and 1mg/kg Ipilimumab | Part E3: 1mg/kg Nivolumab and 3mg/kg Ipilimumab | Part E4: 1mg/kg Nivolumab and 3mg/kg Ipilimumab
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 5 years
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. All-Cause Mortality includes all deaths collected on the study. Ineligible patients are excluded from reporting of adverse events.
Groups:
- Part D: 3mg/kg Nivolumab and 1mg/kg Ipilimumab: Patients with relapsed or refractory neuroblastoma, osteosarcoma, rhabdomyosarcoma, Ewing Sarcoma or Peripheral PNET, Non-Hodgkin Lymphoma, neuroblastoma (MIBG evaluable without RECIST evaluable disease)
Arm/Group | Part A: 3 mg/kg Nivolumab | Part A PK: 3 mg/kg Nivolumab | Part B: 3 mg/kg Nivolumab | Part C: 1mg/kg Nivolumab and 1mg/kg Ipilimumab | Part C: 3mg/kg Nivolumab and 1mg/kg Ipilimumab | Part C PK: 3mg/kg Nivolumab and 1mg/kg Ipilimumab | Part D: 3mg/kg Nivolumab and 1mg/kg Ipilimumab | Part E: 1mg/kg Nivolumab and 3mg/kg Ipilimumab
All-Cause Mortality (participants affected / at risk) | 3/7 | 3/6 | 38/72 | 2/6 | 4/6 | 4/6 | 19/29 | 1/8
Serious Adverse Events (participants affected / at risk) | 6/7 | 6/6 | 70/72 | 4/6 | 6/6 | 5/6 | 26/29 | 7/8
Other Adverse Events (participants affected / at risk) | 7/7 | 6/6 | 72/72 | 6/6 | 6/6 | 6/6 | 29/29 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: 3 mg/kg Nivolumab (N=7) | Part A PK: 3 mg/kg Nivolumab (N=6) | Part B: 3 mg/kg Nivolumab (N=72) | Part C: 1mg/kg Nivolumab and 1mg/kg Ipilimumab (N=6) | Part C: 3mg/kg Nivolumab and 1mg/kg Ipilimumab (N=6) | Part C PK: 3mg/kg Nivolumab and 1mg/kg Ipilimumab (N=6) | Part D: 3mg/kg Nivolumab and 1mg/kg Ipilimumab (N=29) | Part E: 1mg/kg Nivolumab and 3mg/kg Ipilimumab (N=8)
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 4 | 0 | 0 | 0 | 3 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 5 | 1 | 0 | 0 | 2 | 2
Alkaline phosphatase increased (Investigations) | 0 | 0 | 5 | 0 | 0 | 0 | 1 | 0
Allergic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 2 | 25 | 1 | 1 | 2 | 8 | 2
Anorectal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 8 | 0 | 0 | 0 | 4 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 4 | 0 | 2 | 0 | 3 | 1
Autoimmune disorder (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 6 | 0 | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Bronchial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Cardiac disorders - Other, TAMPONADE PHYSIOLOGY (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Catheter related infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cognitive disturbance (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Colonic hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Colonic obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Creatinine increased (Investigations) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Death NOS (General disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 5 | 1 | 0 | 0 | 4 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 6 | 0 | 0 | 0 | 6 | 1
Edema limbs (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye disorders - Other, DECREASED VISION (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye disorders - Other, PRE-SEPTAL CELLULITIS (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye disorders - Other, REDUCED VISION (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye disorders - Other, RIGHT EYE SWELLING (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye disorders - Other, VISION LOSS (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 9 | 0 | 0 | 1 | 1 | 0
Fever (General disorders) | 1 | 0 | 3 | 0 | 1 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
GGT increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gait disturbance (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal disorders - Other, DUODENITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Glucose intolerance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hearing impaired (Ear and labyrinth disorders) | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Hematoma (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hematuria (Renal and urinary disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Hemoglobin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hydrocephalus (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypertension (Vascular disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 3 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0 | 4 | 0 | 0 | 0 | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 8 | 0 | 0 | 1 | 3 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1 | 5 | 2 | 1 | 0 | 4 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0 | 4 | 0 | 0 | 0 | 3 | 1
Hypotension (Vascular disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 5 | 1 | 0 | 0 | 5 | 0
Immune system disorders - Other, GVHD IN THE SETTING OF ALLOTRANSPLANT (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infections and infestations - Other, BLOOD (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infections and infestations - Other, Enterococcus and Pseudomonas pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intestinal stoma leak (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Investigations - Other, CRP INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Investigations - Other, SIADH (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Irregular menstruation (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lipase increased (Investigations) | 0 | 1 | 2 | 0 | 0 | 1 | 4 | 1
Lung infection (Infections and infestations) | 0 | 1 | 4 | 0 | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 3 | 3 | 35 | 1 | 3 | 0 | 12 | 5
Malabsorption (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 1 | 4 | 0 | 0 | 0 | 0 | 0
Multi-organ failure (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal and connective tissue disorder - Other, OSTEOPENIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 0 | 1 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, DISEASE PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, NEUROBLASTOMA PROGRESSI (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, PROGRESSIVE DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 30 | 2 | 3 | 4 | 9 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, PROGRESSIVE DISEASE (EW (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, Progressive Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, due to disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, tumor progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nervous system disorders - Other, Altered mental status (AMS) (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nervous system disorders - Other, Central nervous system dysfunction (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nervous system disorders - Other, SPINAL CORD COMPRESSION - CERVICAL SPINE (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nervous system disorders - Other, SPINAL CORD COMPRESSION - THORACIC SPINE (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 3 | 1 | 26 | 0 | 1 | 1 | 2 | 2
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 0
Obstruction gastric (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 4 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 1 | 0 | 0 | 3 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Paresthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Penile pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Phantom pain (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 3 | 0 | 21 | 0 | 1 | 1 | 4 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 4 | 0 | 0 | 0 | 5 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Psychiatric disorders - Other, AUTISM (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1
Rectal fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal and urinary disorders - Other, Left Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal and urinary disorders - Other, RENAL IMPAIRMENT (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal and urinary disorders - Other, RIGHT HYDRONEPHROSIS (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal calculi (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Respiratory, thoracic and mediastinal disorders - Other, ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Restrictive cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Serum amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin and subcutaneous tissue disorders - Other, CYSTIC ACNE RASH (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Surgical and medical procedures - Other, NEPHROSTOMY (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Surgical and medical procedures - Other, SIGMOID LOOP COLOSTOMY (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Surgical and medical procedures - Other, ULTRASOUND GUIDED CATHETER LUMBAR PLEXUS NERVE BLOCK (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Thromboembolic event (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 11 | 0 | 0 | 0 | 1 | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 4 | 0 | 0 | 1 | 1 | 2
Urine output decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vaginal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vasovagal reaction (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 6 | 0 | 0 | 1 | 0 | 1
Weight gain (Investigations) | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0
Weight loss (Investigations) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
White blood cell decreased (Investigations) | 1 | 2 | 19 | 0 | 1 | 1 | 3 | 2
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: 3 mg/kg Nivolumab (N=7) | Part A PK: 3 mg/kg Nivolumab (N=6) | Part B: 3 mg/kg Nivolumab (N=72) | Part C: 1mg/kg Nivolumab and 1mg/kg Ipilimumab (N=6) | Part C: 3mg/kg Nivolumab and 1mg/kg Ipilimumab (N=6) | Part C PK: 3mg/kg Nivolumab and 1mg/kg Ipilimumab (N=6) | Part D: 3mg/kg Nivolumab and 1mg/kg Ipilimumab (N=29) | Part E: 1mg/kg Nivolumab and 3mg/kg Ipilimumab (N=8)
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 6 | 3
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 22 | 1 | 2 | 1 | 8 | 6
Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 10 | 0 | 0 | 0 | 6 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 3 | 0 | 0 | 1 | 2 | 0
Agitation (Psychiatric disorders) | 0 | 2 | 2 | 0 | 0 | 0 | 2 | 2
Akathisia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 3 | 2 | 34 | 3 | 3 | 2 | 11 | 4
Alkaline phosphatase increased (Investigations) | 3 | 0 | 16 | 2 | 2 | 1 | 6 | 2
Alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Allergic reaction (Immune system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 6 | 2 | 0 | 1 | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 1 | 24 | 1 | 0 | 2 | 10 | 2
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 6 | 6 | 62 | 5 | 6 | 6 | 20 | 6
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 3 | 4 | 28 | 1 | 4 | 2 | 17 | 5
Anxiety (Psychiatric disorders) | 3 | 1 | 18 | 2 | 2 | 1 | 14 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 6 | 0 | 3 | 0 | 2 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 5 | 3 | 36 | 3 | 3 | 4 | 10 | 6
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 0 | 1 | 0 | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 22 | 1 | 2 | 1 | 11 | 4
Bladder spasm (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Bloating (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Blood and lymphatic system disorders - Other, CRP ELEVATED (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood and lymphatic system disorders - Other, LEFT INGUINAL LYMPHADENOPATHY (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood and lymphatic system disorders - Other, MACROCYTOSIS (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 11 | 0 | 1 | 0 | 4 | 2
Blurred vision (Eye disorders) | 0 | 0 | 4 | 1 | 1 | 0 | 5 | 1
Bone marrow hypocellular (Blood and lymphatic system disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 5 | 1 | 0 | 0 | 1 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 1 | 1 | 8 | 0 | 0 | 1 | 3 | 0
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Burn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
CPK increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiac disorders - Other, BENIGN CARDIAC MURMUR (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiac disorders - Other, ECTOPIC ATRIAL RHYTHM (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardiac disorders - Other, HYPERTROPHIC CARDIOMYOPATHY (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiac disorders - Other, RIGHT ATRIAL HYPERTROPHY (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac troponin I increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0 | 0 | 2 | 0 | 0
Chills (General disorders) | 2 | 0 | 5 | 0 | 1 | 1 | 6 | 2
Cholesterol high (Investigations) | 0 | 0 | 2 | 0 | 1 | 0 | 2 | 1
Cognitive disturbance (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Colonic obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Concentration impairment (Nervous system disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Conduction disorder (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Confusion (Psychiatric disorders) | 0 | 1 | 3 | 0 | 0 | 2 | 2 | 1
Conjunctivitis (Eye disorders) | 0 | 0 | 3 | 0 | 1 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 6 | 28 | 2 | 3 | 2 | 14 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 36 | 3 | 3 | 2 | 15 | 4
Creatinine increased (Investigations) | 2 | 1 | 20 | 3 | 1 | 2 | 9 | 3
Cushingoid (Endocrine disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 5 | 1 | 0 | 0 | 5 | 1
Delayed puberty (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 7 | 0 | 0 | 0 | 2 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Depression (Psychiatric disorders) | 1 | 1 | 12 | 0 | 2 | 1 | 6 | 2
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 | 0 | 3 | 0 | 0 | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 1 | 17 | 1 | 0 | 1 | 8 | 4
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 7 | 0 | 0 | 0 | 1 | 2
Dry eye (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 6 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 8 | 2 | 0 | 0 | 5 | 1
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 3 | 0 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 13 | 0 | 1 | 0 | 4 | 4
Ear and labyrinth disorders - Other, EAR INFECTION (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Edema face (General disorders) | 0 | 1 | 4 | 0 | 0 | 0 | 0 | 1
Edema limbs (General disorders) | 2 | 0 | 8 | 0 | 1 | 1 | 7 | 3
Edema trunk (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ejaculation disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 0 | 5 | 0 | 0 | 0 | 3 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Endocrine disorders - Other, ASYMPTOMATIC TSH ELEVATION (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Endocrine disorders - Other, ELEVATED T3 (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Endocrine disorders - Other, ELEVATED TSH (Endocrine disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Endocrine disorders - Other, TSH ELEVATION (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Endocrine disorders - Other, TSH decreased (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Endocrine disorders - Other, thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 8 | 0 | 1 | 0 | 3 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Esophageal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Esophagitis (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0
Euphoria (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
External ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye disorders - Other, ANISOCORIA (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye disorders - Other, ASTIGMATISM (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye disorders - Other, ASYMMETRIC PUPILS (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye disorders - Other, CRUSTY EYES (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye disorders - Other, DIPLOPIA (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye disorders - Other, EYE DISCHARGE (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye disorders - Other, Epicleritis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye disorders - Other, HORNER'S SYNDROME (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye disorders - Other, LEFT ORBIT RECONSTRUCTION (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye disorders - Other, MYOPIA (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye disorders - Other, PAIN, PHOTOPHOBIA AND LID SWELLING OF OD) (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye disorders - Other, PTOSIS (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye disorders - Other, REFRACTIVE ERROR REQUIRING GLASSES (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye disorders - Other, VISION BLACK OUTS (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye disorders - Other, VISUAL IMPAIREMENT (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye pain (Eye disorders) | 1 | 0 | 3 | 1 | 0 | 0 | 2 | 0
Eyelid function disorder (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Facial nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Facial pain (General disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Fatigue (General disorders) | 4 | 4 | 48 | 2 | 4 | 3 | 20 | 8
Fecal incontinence (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 2 | 0
Fever (General disorders) | 2 | 4 | 33 | 2 | 3 | 2 | 14 | 3
Fibrinogen decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 5 | 0 | 1 | 0 | 2 | 1
Flashing lights (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 3 | 0
Floaters (Eye disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Flu like symptoms (General disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 1
Flushing (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0
GGT increased (Investigations) | 1 | 0 | 5 | 1 | 0 | 1 | 0 | 1
Gait disturbance (General disorders) | 3 | 2 | 9 | 1 | 0 | 1 | 5 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 4 | 0 | 0 | 0 | 4 | 1
Gastrointestinal disorders - Other, ABDOMINAL CRAMPING (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal disorders - Other, BURPING (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal disorders - Other, HEARTBURN (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal disorders - Other, INCREASED ORAL SECRETIONS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal disorders - Other, LOOSE TEETH (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal disorders - Other, MOUTH SORE (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal disorders - Other, ORAL PLAQUES (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal disorders - Other, THRUSH (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal disorders - Other, TOOTH SENSITIVITY (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
General disorders and administration site conditions - Other, DECREASED FUNCTIONAL MOBILITY/ACTIVITY (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
General disorders and administration site conditions - Other, GUM SWELLING, LOWER LEFT SIDE (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
General disorders and administration site conditions - Other, HEAD ABRASION (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 6 | 0 | 1 | 0 | 6 | 1
Genital edema (Reproductive system and breast disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gynecomastia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hallucinations (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 3 | 1 | 26 | 4 | 4 | 2 | 11 | 3
Hearing impaired (Ear and labyrinth disorders) | 1 | 1 | 3 | 0 | 1 | 0 | 4 | 1
Heart failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hematuria (Renal and urinary disorders) | 5 | 1 | 15 | 0 | 0 | 1 | 5 | 3
Hemoglobin increased (Investigations) | 2 | 0 | 2 | 0 | 0 | 0 | 2 | 0
Hemoglobinuria (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Hot flashes (Vascular disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1 | 8 | 0 | 0 | 1 | 4 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 3 | 29 | 3 | 3 | 3 | 11 | 7
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 | 13 | 0 | 0 | 0 | 5 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 1 | 13 | 1 | 2 | 0 | 4 | 0
Hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 8 | 0 | 1 | 0 | 3 | 0
Hyperparathyroidism (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypersomnia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 4 | 3 | 17 | 2 | 1 | 1 | 13 | 2
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 8 | 0 | 0 | 0 | 2 | 2
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 0 | 4 | 0 | 0 | 1 | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 4 | 43 | 3 | 3 | 5 | 14 | 6
Hypocalcemia (Metabolism and nutrition disorders) | 4 | 3 | 36 | 3 | 3 | 2 | 9 | 6
Hypoglossal nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 1 | 10 | 0 | 0 | 0 | 2 | 2
Hypohidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 3 | 3 | 22 | 3 | 2 | 1 | 10 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 25 | 0 | 1 | 1 | 7 | 4
Hyponatremia (Metabolism and nutrition disorders) | 2 | 4 | 40 | 4 | 2 | 3 | 13 | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 3 | 28 | 2 | 1 | 2 | 10 | 3
Hypotension (Vascular disorders) | 1 | 0 | 14 | 0 | 1 | 0 | 8 | 3
Hypothermia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 3 | 1 | 19 | 0 | 2 | 2 | 9 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 3 | 0 | 0 | 0 | 0 | 1
INR increased (Investigations) | 0 | 0 | 6 | 0 | 1 | 0 | 4 | 2
Immune system disorders - Other, HYPOGAMMAGLOBULINEMIA (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infections and infestations - Other, C. DIFFICILE (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infections and infestations - Other, BACTEREMIA (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infections and infestations - Other, C.DIFF (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infections and infestations - Other, E.COLI (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infections and infestations - Other, ESR ELEVATED (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infections and infestations - Other, INFLUENZA B (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infections and infestations - Other, KLEBSIELLA BACTEREMIA (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infections and infestations - Other, POS blood CX (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infections and infestations - Other, RESPIRATORY SYNCYTIAL VIRUS RNA (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infections and infestations - Other, RHINORREA (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infections and infestations - Other, RHINOVIRUS/ENTEROVIRUS (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infections and infestations - Other, STERILE ABCESS (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infections and infestations - Other, Strep throat (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infections and infestations - Other, THRUSH (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infections and infestations - Other, UPPER RESPIRATORY INFECTION (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 4 | 0 | 1 | 0 | 1 | 1
Injection site reaction (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Injury, poisoning and procedural complications - Other, Forehead laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 15 | 0 | 0 | 2 | 8 | 3
Intestinal stoma leak (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Investigations - Other, (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Investigations - Other, BICARBONATE LOW (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Investigations - Other, (ELEVATED CRP) (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, ALT DECREASED (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Investigations - Other, AMYLASE DECREASED (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, AMYLASE, DECREASED (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Investigations - Other, ANION GAP INCREASED (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Investigations - Other, Amylase Increase (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, BICARB INCREASED (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Investigations - Other, BICARBONATE (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Investigations - Other, BICARBONATE SERUM LOW (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Investigations - Other, BLOOD LDH INCREASED (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, BUN DECREASED (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Investigations - Other, BUN HIGH (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, BUN INCREASED (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Investigations - Other, C REACTIVE PROTEIN (Investigations) | 0 | 0 | 6 | 0 | 0 | 0 | 1 | 0
Investigations - Other, C REACTIVE PROTEIN ELEVATED (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Investigations - Other, C REACTIVE PROTEIN INCREASED (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Investigations - Other, C-REACTIVE PROT (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, C-REACTIVE PROTEIN (Investigations) | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0
Investigations - Other, C-REACTIVE PROTEIN ELEVATED (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Investigations - Other, C-REACTIVE PROTEIN INCREASED (Investigations) | 0 | 0 | 8 | 0 | 0 | 0 | 4 | 0
Investigations - Other, C-REATIVE PROTEIN INCREASED (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, C-Reactive Prot. (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, C-Reactive prot. increase (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, C-Reactive protein (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, C-Reactive protein increase (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, C02 LOW (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Investigations - Other, CARBON DIOXIDE (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, CHLORIDE (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, CHLORIDE DECREASED (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, CHLORIDE INCREASED (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, CHLORIDE LOW (Investigations) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Investigations - Other, CO2 LOW (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Investigations - Other, CREATININE DECREASED (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Investigations - Other, CREATININE, DECREASED (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Investigations - Other, CRP (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, CRP ELEVATED (Investigations) | 0 | 0 | 7 | 0 | 0 | 0 | 0 | 0
Investigations - Other, CRP HIGH (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, CRP INCREASE (Investigations) | 0 | 0 | 2 | 0 | 0 | 3 | 0 | 0
Investigations - Other, CRP INCREASED (Investigations) | 0 | 1 | 16 | 1 | 0 | 1 | 5 | 0
Investigations - Other, CRP increase (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Investigations - Other, CRP increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Investigations - Other, CRP, ELEVATED (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Investigations - Other, DECREASE CHLORIDE (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Investigations - Other, DECREASED BICARBONATE (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Investigations - Other, ELEVATED BUN (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, ELEVATED C REACTIVE PROTEIN (Investigations) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Investigations - Other, ELEVATED C-REACTIVE PROTEIN (Investigations) | 2 | 0 | 6 | 1 | 0 | 0 | 3 | 0
Investigations - Other, ELEVATED C-REATIVE PROTEIN (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, ELEVATED CRP (Investigations) | 1 | 2 | 9 | 1 | 1 | 0 | 8 | 0
Investigations - Other, ELEVATED ESR (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, ELEVATED LDH (Investigations) | 2 | 1 | 1 | 0 | 0 | 1 | 1 | 0
Investigations - Other, EOSINOPHIL COUNT INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Investigations - Other, ESR INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Investigations - Other, FREE T4 LOW (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Investigations - Other, GLUCOSE IN URINE (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, HIGH CRP VALUE (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, HYPERBILIRUBINEMIA (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Investigations - Other, HYPERCHLOREMIA (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, HYPERPHOSPHATEMIA (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Investigations - Other, HYPOCHLOREMIA (Investigations) | 2 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Investigations - Other, HYPOURICEMIA (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, Hypochloremia (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Investigations - Other, INCREASED ANION GAP (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Investigations - Other, INCREASED C REACTIVE PROTEIN (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Investigations - Other, INCREASED C-REACTIVE PROTEIN (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, INCREASED CARBON DIOXIDE LEVEL (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Investigations - Other, INCREASED CHLORIDE (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, INCREASED CRP (Investigations) | 1 | 0 | 3 | 0 | 0 | 0 | 4 | 0
Investigations - Other, INCREASED TSH (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, INCREASED WBC (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Investigations - Other, INFLUENZA (A) (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, Increased Bands (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Investigations - Other, LDH ELEVATED (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, LDH INCREASE (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, LDH INCREASED (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Investigations - Other, LI[PASE, DECREASED (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Investigations - Other, LOW BICARB (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, LOW BICARBONATE (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Investigations - Other, LOW C-REACTIVE PROTEIN (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Investigations - Other, LOW CO2 (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, LOW VITAMIN D (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Investigations - Other, LYMPHOPENIA (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Investigations - Other, MCHC DECREASED (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, NEUROPHILA (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, NON FASTING GLUCOSE (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Investigations - Other, PHOSPHORUS INCREASED (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, PLATELET COUNT INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Investigations - Other, PT PROLONGED (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, PTT SHORTENED (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Investigations - Other, RIGHT LOWER BACK PRESSURE (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, SERUM OSMOLARITY DECEASE (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, SERUM PROTEIN DECREASED (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Investigations - Other, TINGLING IN HANDS/NEURO PAIN (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, TOTAL PROTEIN (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, TOTAL PROTEIN DECREASED (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, TSH ELEVATED (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, TSH HIGH (Investigations) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Investigations - Other, TSH INCREASED (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, TSH LOW (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, VIT D DEFICIENCY (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Investigations - Other, VITAMIN D DEFICIENCY (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Investigations - Other, Vitamin D decrease (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Investigations - Other, lipase increase (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Irritability (General disorders) | 1 | 2 | 5 | 1 | 0 | 1 | 4 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 2 | 0 | 6 | 2 | 0 | 0 | 8 | 0
Joint range of motion decreased cervical spine (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Kyphosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Lip infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lip pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lipase increased (Investigations) | 0 | 0 | 5 | 0 | 1 | 2 | 5 | 1
Localized edema (General disorders) | 0 | 0 | 3 | 2 | 0 | 1 | 5 | 0
Lung infection (Infections and infestations) | 1 | 0 | 3 | 0 | 0 | 0 | 2 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphedema (Vascular disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 5 | 3 | 37 | 3 | 2 | 2 | 17 | 7
Lymphocyte count increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 5 | 0 | 1 | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Metabolism and nutrition disorders - Other, BICARBONATE DECREASE (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Metabolism and nutrition disorders - Other, CRP ELEVATED (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Metabolism and nutrition disorders - Other, DECREASED CARBON DIOXIDE (CO2), (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Metabolism and nutrition disorders - Other, DECREASED PROTEIN (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Metabolism and nutrition disorders - Other, ELEVATED BICARBONATE (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Metabolism and nutrition disorders - Other, ELEVATED TSH (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Metabolism and nutrition disorders - Other, HYPOCHLOREMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mitral valve disease (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Movements involuntary (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal infection (Infections and infestations) | 0 | 1 | 3 | 0 | 0 | 1 | 2 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 5 | 0 | 0 | 1 | 3 | 1
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 2 | 0 | 0 | 1 | 0
Musculoskeletal and connective tissue disorder - Other, AMBULATES WITH LIMP (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal and connective tissue disorder - Other, ANKLE PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, CHEST WALL MASS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, CRACKING/SQUEAKING (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal and connective tissue disorder - Other, DECONDITIONING (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, HAND AND LEG CRAMPING (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, HEAD - LARGE INDENTION IN OCCIPITAL SCALP (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal and connective tissue disorder - Other, HIP PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, LIMBS MUSCLE CRAMPING (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Musculoskeletal and connective tissue disorder - Other, SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, SWELLING (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, SWELLING OF LT MID BACK (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 5 | 0 | 2 | 1 | 3 | 2
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 16 | 1 | 1 | 0 | 7 | 3
Nausea (Gastrointestinal disorders) | 4 | 4 | 36 | 1 | 1 | 2 | 15 | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 4 | 0 | 1 | 0 | 2 | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, INTRATUMOR HEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, TUMOR SWELLING, LEFT FO (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, TUMOR SWELLING: LEFT TH (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nervous system disorders - Other, DECREASED REFLEXES (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nervous system disorders - Other, HYPERALGESIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nervous system disorders - Other, LIGHT-HEADED (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nervous system disorders - Other, MENTAL STATUS CHANGES (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nervous system disorders - Other, PARAPLEGIC IN LEGS (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nervous system disorders - Other, SPINAL CORD COMPRESSION (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nervous system disorders - Other, WEARS GLASSES (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Neutrophil count decreased (Investigations) | 3 | 4 | 23 | 2 | 3 | 0 | 8 | 4
Non-cardiac chest pain (General disorders) | 0 | 2 | 10 | 1 | 2 | 0 | 7 | 4
Nystagmus (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Obstruction gastric (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oculomotor nerve disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Optic nerve disorder (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral hemorrhage (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1 | 4 | 0 | 0 | 0 | 2 | 1
Otitis media (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Ovulation pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 1 | 3 | 19 | 1 | 1 | 1 | 6 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 4 | 26 | 3 | 1 | 0 | 15 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pancreatic enzymes decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Paresthesia (Nervous system disorders) | 0 | 0 | 5 | 1 | 1 | 1 | 2 | 2
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Paroxysmal atrial tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Penile pain (Reproductive system and breast disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 6 | 2 | 1 | 0 | 3 | 0
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Periorbital edema (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 3 | 9 | 0 | 0 | 1 | 5 | 2
Personality change (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Phantom pain (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Photophobia (Eye disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 4 | 4 | 37 | 3 | 3 | 2 | 10 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 11 | 2 | 1 | 0 | 10 | 1
Pleural hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 3 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 6 | 1 | 0 | 0 | 4 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 20 | 1 | 5 | 4 | 11 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 2 | 13 | 0 | 0 | 0 | 4 | 2
Psychiatric disorders - Other, ADHD (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Psychiatric disorders - Other, DYSPHORIA (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Psychiatric disorders - Other, EXCORIATION/SKIN PICKING (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Psychiatric disorders - Other, HX OF ADD (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Psychiatric disorders - Other, SPEECH/LANGUAGE DISORDER (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Radiculitis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 5 | 2 | 1 | 0 | 1 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 2 | 12 | 3 | 2 | 0 | 3 | 1
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Rectal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal and urinary disorders - Other, 1 + KETONES IN URINE (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal and urinary disorders - Other, DYSURIA (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal and urinary disorders - Other, FANCONI PROXIMAL TUBULE RENAL DISEASE. (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal and urinary disorders - Other, GLUCOSURIA (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Renal and urinary disorders - Other, HYDRONEPHROSIS (Renal and urinary disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Renal and urinary disorders - Other, HYDRONEPHROSIS W/ PELVOCALICETASIS (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Renal and urinary disorders - Other, HYDRONEPHROSIS/URINARY CATHETERIZATION (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Renal and urinary disorders - Other, KETONURIA (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal and urinary disorders - Other, MUCOUS IN URINE (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal and urinary disorders - Other, Nephrostomy tube bleeding (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal and urinary disorders - Other, OLIGURIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal and urinary disorders - Other, TRACE URINE PROTEIN (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal and urinary disorders - Other, URINARY HESITANCY (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal and urinary disorders - Other, URINE GLUCOSE (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Renal and urinary disorders - Other, URINE MUCUS (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal and urinary disorders - Other, URINE RBCS (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal and urinary disorders - Other, URINE URBILINOGEN (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal and urinary disorders - Other, URINE WBCS (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Reproductive system and breast disorders - Other, (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Reproductive system and breast disorders - Other, PRIMARY OVARIAN FAILURE (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other, BILATERAL AIRSPACE DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, BRADYPNEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, BURNING NOSTRILS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other, DRY, SCRATCHY THROAT (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, HEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other, INCREASED WORK OF BREATHING (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, INTERMITTENT HEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other, RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, RHINORRHEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 1 | 0 | 2 | 0
Respiratory, thoracic and mediastinal disorders - Other, RUNNY NOSE (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, TACHYPNEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 7 | 0 | 0 | 0 | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other, Tachypnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Restlessness (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Retinopathy (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinitis infective (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Scleral disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Scrotal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Serum amylase increased (Investigations) | 0 | 0 | 5 | 1 | 2 | 3 | 1 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 3 | 1 | 0 | 0 | 4 | 1
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Sinus tachycardia (Cardiac disorders) | 5 | 3 | 28 | 2 | 2 | 3 | 19 | 3
Sinusitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 3 | 0
Skin and subcutaneous tissue disorders - Other, ABRASION TO FACE (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin and subcutaneous tissue disorders - Other, ABRASIONS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, BLISTERS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, BUG BITES (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, BUG BITES ON SCALP. (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin and subcutaneous tissue disorders - Other, CAFE AU LAIT ON ABDOMEN (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, CHAPPED LIPS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, CIRCULAR, FLAT AREA WITH REDNESS ON BACK (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, CONTACT DERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin and subcutaneous tissue disorders - Other, DARK UNDER-EYE CIRCLES (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin and subcutaneous tissue disorders - Other, DERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, DESQUAMATION (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, DIAPER DERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, DRY LIPS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, ERYTHEMA ON R ANTECUBITAL (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, ERYTHEMA RIGHT HIP (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, ERYTHEMATOUS MACULAR RASH (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, ERYTHEMATOUS RASH (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, ERYTHEMATOUS SPOT ON PENIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, ERYTHEME AROUND EYELIDS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, EXCORIATIONS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, FAINT ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, FEW SCATTERED INSECT BITES ON FOREHEAD. (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, INSECT BITES (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, ITCHING (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, LESION ON UPPER LIP (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, MILD DIFFUSE REDNESS ARMS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, MILD ERYTHEMIA (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, NEVUS FLAMMEUS ON R FACE & OROPHARYNX (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, NEVUS LESIONS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, NON-RAISED, NON-PRURITIC RASH TO CHEEKS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin and subcutaneous tissue disorders - Other, ORAL THRUSH (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin and subcutaneous tissue disorders - Other, PAPULAR RASH (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin and subcutaneous tissue disorders - Other, PIMPLES (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, RASH (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin and subcutaneous tissue disorders - Other, SEVERAL PETECHIAE. (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, SKIN LESION UNDER NOSE (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, SLIGHT ERYTHEMA OF SKIN OVERLYING RIGHT AXILLARY MAS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin and subcutaneous tissue disorders - Other, STASIS DERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin and subcutaneous tissue disorders - Other, STRIAE (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin and subcutaneous tissue disorders - Other, TINY PAPULES ON SHOULDER AND UPPER ABDOMEN (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, UNKNOWN SKIN LESIONS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin and subcutaneous tissue disorders - Other, WARTS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin and subcutaneous tissue disorders - Other, WHITE BLOTCHES ON ABDOMEN (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 5 | 0 | 0 | 0 | 3 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 1 | 3 | 0 | 0 | 0 | 1 | 0
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 2 | 6 | 1 | 0 | 1 | 3 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 8 | 0 | 1 | 1 | 6 | 2
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Stomach pain (Gastrointestinal disorders) | 0 | 1 | 5 | 0 | 1 | 1 | 5 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thromboembolic event (Vascular disorders) | 0 | 0 | 4 | 0 | 1 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Tooth discoloration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Tricuspid valve disease (Cardiac disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Trigeminal nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 9 | 2 | 0 | 1 | 4 | 1
Upper respiratory infection (Infections and infestations) | 0 | 0 | 8 | 1 | 0 | 0 | 5 | 1
Urinary frequency (Renal and urinary disorders) | 0 | 0 | 5 | 0 | 0 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 5 | 0 | 0 | 1 | 4 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 9 | 0 | 0 | 1 | 2 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 5 | 0 | 0 | 1 | 0 | 2
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Urinary urgency (Renal and urinary disorders) | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 2
Urine discoloration (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Uveitis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vaginal pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vascular disorders - Other, (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3 | 30 | 2 | 1 | 2 | 17 | 4
Watering eyes (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Weight gain (Investigations) | 2 | 0 | 3 | 1 | 0 | 1 | 1 | 2
Weight loss (Investigations) | 1 | 3 | 14 | 3 | 2 | 2 | 10 | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 6 | 0 | 1 | 0 | 4 | 0
White blood cell decreased (Investigations) | 4 | 4 | 40 | 2 | 3 | 1 | 11 | 4
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-30): https://cdn.clinicaltrials.gov/large-docs/58/NCT02304458/Prot_SAP_000.pdf